CLINICAL TRIAL: NCT04367584
Title: Comparison of Malassezia Spp Proportions in Inflammatory and Non Inflammatory Facial Acne Vulgaris Lesions
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Agassi Suseno Sutarjo, SpKK, Principal investigator, Indonesia University
Other Study IDs: 18-09-1019
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Acne Vulgaris
Keywords: Acne lesion, Malassezia spp, skin microbiome, pruritus
MeSH Terms: conditions — Acne Vulgaris; Pruritus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with inflammatory AV lesions: Clinical examination Laboratory examination (follicular content of acne lesions were obtained for fungal microscopic examination and fungal culture)
  Interventions: Other: Clinical and laboratory examination
- Subjects with non inflammatory AV lesions: Clinical examination Laboratory examination (follicular content of acne lesions were obtained for fungal microscopic examination and fungal culture)
  Interventions: Other: Clinical and laboratory examination

INTERVENTIONS:
Other: Clinical and laboratory examination — Clinical and laboratory examination (follicular content of acne lesions were obtained for fungal microscopic examination and fungal culture)

SUMMARY:
Acne vulgaris (AV) is a common inflammatory condition involving pilosebaceous unit. The pathogenesis of acne is multifactorial and skin microbiome is considered to be one of the key factors that aggravate inflammation. Malassezia spp is normal flora on the skin and several studies have reported its corelation with inflammatory AV lesion.

Malassezia have higher lipase activity compared to Propionibacterium acnes which triggers an increase in free fatty acid and glycerol, the chemotactic factors towards neutrophils and inducing inflammation in AV. Malassezia folliculitis (MF) is sometimes confused with and may present together with AV. Pruritus usually presents in MF but some studies also reported itching as common symptom in AV.

The objectives of this study were to identify the presence and the distribution of Malassezia spp. in facial AV lesions, to compare the distribution of Malassezia spp. between inflammatory and non-inflammatory lesions and to identify the association between Malassezia spp in acne lesions and pruritus symptom.

DETAILED DESCRIPTION:
This study used cross sectional design study.

Subjects with eligible criteria were included. Subjects were divided into subjects with inflammatory lesions and subjects with non inflammatory lesions.

Physical examination consisted of assesment of AV severity (using Lehman criteria) and presence of pruritus based on visual analog scale. Clinical documetations were taken.

Follicular content of four inflammatory lesions or four non inflammatory lesions were collected for microscopic examination with KOH solution and fungal culture examination (using CHROMagar Malassezia, Dextrose Saboraud agar (DSA), and Tween 60-esculin agar).

The presence of Malassezia spp and its spore load in both groups were assesed and analyzed for its corelation with AV severity and presence of pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with age of 15-49 years with AV and the presence of at least four inflammatory and four non-inflammatory lesions

Exclusion Criteria:

* Subjects with prior topical retinoid acid or topical antifungal medication within the past two weeks, systemic antibiotic or antifungal use within the past month, and corticosteroid use within the past six months

Ages: 15 Years to 49 Years | Sex: All
Age Groups: Child, Adult
Study Population: Subjects with age of 15-49 years and the presence of at least four inflammatory and four non-inflammatory acne lesions at Dermatology-Venereology outpatient clinic in a tertiary hospital in Indonesia between October to November 2018.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Malassezia spp. from culture examination | Sample collected during subjects enrollment
  Proportion of Malassezia spp. from culture of inflammatory and non-inflammatory facial AV lesions

SECONDARY OUTCOMES:
Proportion of fungal spore load based on microscopic examination | Sample collected during subjects enrollment
  Proportion of fungal spore load of inflammatory and non-inflammatory facial AV lesions based on microscopic examination graded using Jacinto Jamora criteria
Presence and severity of pruritus | Data collected during subjects enrollment
  Presence and severity of pruritus graded using visual analog scale in correlation with the presence of Malassezia spp and its spore load

CONTACTS AND LOCATIONS:
Overall Officials: Agassi Suseno Sutarjo, MD, Principal Investigator — Department of Dermatology and Venereology, Tarakan General Hospital, Indonesia
Locations (1):
- Dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided